CLINICAL TRIAL: NCT00884455
Title: Alpha-1 Foundation DNA and Tissue Bank
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: Alpha-1 Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201500842 AATD Tissue Bank
Record Dates: First submitted 2009-04-17; First posted 2009-04-20 (Estimated); Last update posted 2026-01-15 (Actual); Status verified 2025-08

CONDITIONS: Alpha 1 Antitrypsin Deficiency
Keywords: tissue banking, research
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, liver and lung
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a long-term follow-up banking protocol that collects medical information and tissue (blood, liver and lung) samples for future research; use of data and samples for research purposes is overseen by the Tissue Bank Advisory Committee; the purpose of the Bank is to further research on alpha-1 antitrypsin deficiency.

DETAILED DESCRIPTION:
Subject participation includes completion of informed consent, medical questionnaire, and email authorization. Subjects may provide a blood sample for alpha-1 antitrypsin genotype, phenotype and level. Lung and liver tissue may also be provided if available. Subjects may be contacted no more often than annually for updated information.

This project has a certificate of confidentiality from NIH.

ELIGIBILITY:
Inclusion Criteria:

* all interested individuals may enroll

Exclusion Criteria:

* there are no exclusion criteria

Ages: 0 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: subjects with alpha-1-antitrypsin deficiency, carriers of deficient alleles and interested individuals
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2002-12 (Actual); Primary Completion 2032-06-10 (Estimated); Study Completion 2033-06-10 (Estimated)

PRIMARY OUTCOMES:
Data and tissue samples | The total number of tissue samples received and used for research are tracked annually.
  At the end of 15 years the tissue and data sample usage will be analyzed to determine continuation of the project. Each year the investigator provides a summary to the Alpha-1 Foundation.

CONTACTS AND LOCATIONS:
Overall Officials: Karina Serban, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

REFERENCES:
- [Result] Tonelli AR, Rouhani F, Li N, Schreck P, Brantly ML. Alpha-1-antitrypsin augmentation therapy in deficient individuals enrolled in the Alpha-1 Foundation DNA and Tissue Bank. Int J Chron Obstruct Pulmon Dis. 2009;4:443-52. doi: 10.2147/copd.s8577. Epub 2009 Dec 29. PMID 20054436
- [Result] Clark VC, Dhanasekaran R, Brantly M, Rouhani F, Schreck P, Nelson DR. Liver test results do not identify liver disease in adults with alpha(1)-antitrypsin deficiency. Clin Gastroenterol Hepatol. 2012 Nov;10(11):1278-83. doi: 10.1016/j.cgh.2012.07.007. Epub 2012 Jul 24. PMID 22835581